CLINICAL TRIAL: NCT00921284
Title: Closed-Loop Delivery of Propofol and Remifentanil: Sparing Effect of Dexmedetomidine
Brief Title: Influence of Dexmedetomidine on a Closed-Loop Anesthesia System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008/41
Record Dates: First submitted 2009-06-13; First posted 2009-06-16 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and a placebo
  Interventions: Drug: NaCl 9/00
- dexmedetomidine (Experimental): patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and dexmedetomidine
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: NaCl 9/00 — Same volume as in the dexmedetomidine group
  Arms: Placebo
Drug: dexmedetomidine — 1 mcg/kg administered in 10 minutes followed by a continuous infusion of 0,5 mcg/kg/hr
  Arms: dexmedetomidine

SUMMARY:
The main objective if to evaluate the sparing effect of dexmedetomidine on the doses of propofol and remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* male patients scheduled for a general anesthesia

Exclusion Criteria:

* age lower than 18 years
* allergy to propofol, or to soja or to peanuts, or to sufentanil, to remifentanil, or to morphine,or to a myorelaxant or to an excipient,
* hypersensibility to sufentanil, or to remifentanil, or to other derivate of fentanyl,
* history of central nervous system disease,
* patients receiving a psychotropic treatment or an agonist-antagonist opiate,
* hypovolemic patients,
* patients receiving a cardio-vascular treatment,
* expected bleeding surgical procedure,
* simultaneous general and loco-regional anesthesia,
* severe hepatic insufficiency.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
administered doses of propofol and of remifentanil during anesthesia | end of anesthesia

SECONDARY OUTCOMES:
delay before recovery | at the end of anesthesia
hemodynamic abnormalities requiring a treatment | end of anesthesia
postoperative morphine requirement | Third post-anesthetic hour
explicit memorisation | Second postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (1):
- Hôpital Foch, Suresnes, France